CLINICAL TRIAL: NCT02875548
Title: Tazemetostat Rollover Study (TRuST): An Open-Label, Rollover Study
Brief Title: A Study to Assess Long-term Safety of Tazemetostat in Adult Participants of All Ages With Any Disease Treated With Tazemetostat in a Previous Clinical Study
Acronym: TRuST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-501; 2015-004984-35 (EudraCT Number); 2023-510553-41-00 (EU CTIS Number)
Record Dates: First submitted 2016-08-05; First posted 2016-08-23 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Synovial Sarcoma; Epitheliod Sarcoma (ES); Mesothelioma; Advanced Solid Tumors; Renal Medullary Carcinoma; Non-Hodgkin Lymphoma (NHL)
Keywords: Epizyme; Tazverik; Tazemetostat (EPZ-6438)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Sarcoma, Synovial; Mesothelioma; Lymphoma, Non-Hodgkin | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Tazemetostat (Experimental): Participants will continue to receive the same tazemetostat dose and schedule as specified in their antecedent tazemetostat protocol.
  For participants on combination therapy, the other therapeutic(s) must have been completed in the antecedent study or be provided by a source other than Epizyme if combination treatment is continued in this clinical rollover study.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of enhancer of Zeste homolog 2 (EZH2), a histone-lysine N-methyltransferase enzyme.
  Other Names: EPZ-6438; E7438; IPN60200

SUMMARY:
This study will provide continuing availability to tazemetostat for people that have previously completed participation in a tazemetostat study, either with monotherapy (single drug treatment) or combination therapy.

The aim of the study will be to assess the long-term safety of tezemetostat.

DETAILED DESCRIPTION:
This open-label, multicenter, global study will provide continuing access to tazemetostat therapy for subjects who have completed their participation in a prior tazemetostat study (either with monotherapy or combination therapy)

without unacceptable toxicity, have not had evidence of tumor progression as defined by disease-appropriate standard criteria, and continue to receive clinical benefit from the therapy.

Subjects will receive tazemetostat as dictated in their antecedent study. Visits will be conducted per Standard of Care (SoC) as appropriate in each country and as determined by the Investigator. Subjects will be followed for long-term safety in addition to time to treatment failure (TTF) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet ALL criteria to be eligible for enrollment in this study.
2. Has demonstrated and continues to demonstrate clinical benefit from treatment with tazemetostat.
3. Is currently receiving tazemetostat as either monotherapy or in combination with other approved drug(s) or investigational agent(s) on an Epizyme-sponsored clinical trial or any other clinical trial being conducted with tazemetostat that is not sponsored by Epizyme (including but not limited to, investigator-initiated trials). For subjects on combination therapy, treatment with other therapeutic(s) must have been completed in the antecedent study or will be provided by a source other than Epizyme if combination therapeutics are continued in this study until disease progression, treatment toxicity, subject preference or death, up to approximately 7 years.
4. Has voluntarily provided signed written informed consent and demonstrated willingness and ability to comply with all aspects of the protocol.
5. Has a life expectancy of ≥3 months.
6. Has adequate hematologic, (bone marrow [BM] and coagulation factors), renal, and hepatic function. Subject must remain eligible for continued treatment with tazemetostat according to the eligibility and treatment criteria from the antecedent study

Exclusion Criteria:

Subjects meeting ANY of the following criteria must NOT be enrolled in this study:

1. Has had an interruption of tazemetostat dosing of >14 days from the antecedent clinical study to starting the rollover study unless approved by the Medical Monitor.
2. Has another malignancy other than the one for which they are receiving tazemetostat.

   • Exception: Subject who has been disease-free of a prior malignancy for 5 years or subject with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is eligible.
3. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE v5 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).
4. Has a prior history of T-LBL/T-ALL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Treatment Emergent Adverse Event (TEAEs) | Until end of study an average of 7 years
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention Severity of adverse events experienced by all participants will be evaluated by the Investigator based on the CTCAE, version 5.0.
Duration of Study Drug Exposure | Until end of study an average of 7 years
  The average study drug exposure duration will be reported.

SECONDARY OUTCOMES:
The overall survival (OS) | Until end of study an average of 7 years
  Defined as the interval of time between the date of the first dose of tazemetostat and the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (34):
- United States (11):
  - University of Arizona Cancer Center, Tucson, Arizona
  - California Cancer Associates For Research And Excellence, cCARE, Santa Fe, California
  - Hematology Oncology Associates of the Treasure Coast - Port St. Lucie, Port Saint Lucie, Florida
  - Moffitt, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Central Care Cancer Center, Bolivar, Missouri
  - Astera Cancer Center, East Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - David H. Koch Center for Cancer Care at memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (5):
  - Princess Alexandra Hospital, Alexandra
  - Monash Medical Centre- Monash Campus, Clayton
  - Geelong Hospital, Geelong
  - Peter MacCallum Cancer Institute, Melbourne
  - Monash Health, Monash
- University Hospital (UZ) Leuven, Leuven, Belgium
- France (9):
  - Institut Bergonie, Bordeaux
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHRU de Lile- Hopital Claude Huriez, Lille
  - CHU de Montpellier - Hopital Saint Eloi, Montpellier
  - Hôpital Saint Louis - AP-HP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Rennes- Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Gustave Roussay, Villejuif
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Klinika Endokrynologii Onkologicznej i Medycyny Nuklearnej, Warsaw
- S.P. Grigoreva Institute of Medical Radiology and Oncology of NAMS of Ukraine", Kharkiv, Ukraine
- United Kingdom (5):
  - Beatson, West of Scotland Cancer Centre, Glasgow
  - Oncology and Haematology Clinical Trials Unit, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/